CLINICAL TRIAL: NCT00005408
Title: Reanalysis of CVD Risk Factors Via Likelihood Methods
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4326; R03HL046674 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis

SUMMARY:
To reanalyze data on risk factors for cardiovascular disease (CVD) including total cholesterol and high density lipoprotein (HDL) cholesterol for the subjects in the first, second, and third exams of the NHLBI Twin Study.

DETAILED DESCRIPTION:
BACKGROUND:

The results of these longitudinal analyses yielded new insights on genetic effects affecting CVD risk factors during the aging process.

DESIGN NARRATIVE:

The analyses utilized maximum likelihood estimators of genetic variance which were asymptotically more efficient than the method-of-moments estimators used in previous analyses. The models used incorporated terms to partition the variance in a trait from twin data into either i) additive genetic variance and unshared environmental variance (the AE model), ii) additive genetic variance, dominance genetic variance, and unshared environmental variance (the ADE model), or iii) additive genetic variance, shared environmental variance, and unshared environmental variance (the ACE model). The AE, ADE, and ACE models were fitted separately to data from each of the three exams to obtain a cross-sectional analysis. The investigators also extended these models for use with longitudinal data by incorporating terms to represent the covariance of variance components from different exams.

Two important additional objectives of this study were i) to introduce resistant estimation techniques in twin modeling, which trimmed the effect of outlier data points smoothly, and ii) to carefully study the performance of maximum likelihood and method-of-moments estimators when assumptions of the twin model were violated. The results of these parts of the study should yield a more complete understanding of the relative merits and limitations of twin modeling procedures.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-07; Study Completion 1994-04 (Actual)

REFERENCES:
- [Background] Williams CJ, Wijesiri UW. Lipid data from NHLBI veteran twins: interpreting genetic analyses when model assumptions fail. Genet Epidemiol. 1993;10(6):551-6. doi: 10.1002/gepi.1370100637. PMID 8314059
- [Background] Williams CJ. On the covariance between parameter estimates in models of twin data. Biometrics. 1993 Jun;49(2):557-68. PMID 8369388
- [Background] Wijesiri UW, Williams CJ. Approximate solutions for the maximum-likelihood estimates in models of univariate human twin data. Behav Genet. 1995 May;25(3):211-6. doi: 10.1007/BF02197179. PMID 7598664